CLINICAL TRIAL: NCT06042049
Title: A Phase III Single-Arm Open-Label Study to Evaluate the Safety PK ADA and Anti RSV nAb Following Administration of 2 Doses of Nirsevimab Given 5 to 6 Months Apart in Infants With CHD, CLD, Immunocompromise, Down Syndrome, or Born Pre-Term in Japan
Brief Title: A Study to Assess Safety, Pharmacokinetics Anti-Drug Antibody and Anti-RSV Antibody After 2 Doses of Nirsevimab
Acronym: JUBILUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D5290C00009; 2025-000021-13 (EudraCT Number)
Record Dates: First submitted 2023-07-13; First posted 2023-09-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — nirsevimab

STUDY DESIGN:
Masking Description: No masking is used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEDI8897 (Experimental): Anti-RSV monoclonal antibody
  Interventions: Drug: Nirsevimab

INTERVENTIONS:
Drug: Nirsevimab — Participants in the first year of life will receive the 1st dose of nirsevimab as a single, fixed intramuscular (IM) dose of 50 mg if body weight is <5 kg or 100 mg if body weight is ≥5 kg. A 2nd fixed IM dose of 50 mg if body weight is <5 kg or 100 mg if body weight is ≥5 kg will be administered 5 to 6 months following the 1st dose.
  Other Names: MEDI8897

SUMMARY:
The purpose of this study is to measure the safety, PK, occurrence of ADA to nirsevimab, and anti-RSV neutralizing Ab in Japanese children with certain health conditions or pre-term infants aged ≤12 months.

Study details include

* The study duration is approximately 21 months with a 2-month enrollment period.
* Study intervention is 2 doses administered 5- 6 months apart.
* The study has 5 or 6 site visits and several telephone contacts with a 2 or 4 week interval.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally required authorization obtained from the participant's parent(s)/legally authorized representative(s) before performing any protocol-related procedures, including screening evaluations
2. Japanese infants of ≤12 months of age eligible to receive palivizumab in accordance with national or local guidelines and those who must meet at least one of the following conditions at the time of informed consent.

   1. Immunodeficiency
   2. Chronic Lung Disease
   3. Congenital Heart Disease
   4. Down syndrome
   5. Born pre-term ≤28 wks Gestation age and aged ≤12 months, or born pre-term >28 wks and ≤35 wks Gestation age and aged ≤6 months
3. The participant's parent(s)/legally authorized representative(s) can understand and comply with the requirements of the protocol including follow-up visits as judged by the investigator.
4. The participant is available to complete the follow-up period for approximately 19 months, which will be approximately 1 year after receipt of 2nd dose of nirsevimab

Exclusion Criteria:

1. Requirement for mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure (CPAP), or other mechanical respiratory or cardiac support at the time of enrollment
2. A current, active RSV infection at the time of screening and investigational product administration
3. Any fever (≥100.4°F [≥38.0°C], regardless of route) or acute illness at the time of prior to investigational product administration
4. Any serious concurrent medical condition (except those resulting in an immune deficiency condition), including:

   1. Known renal impairment
   2. Known hepatic dysfunction including known or suspected active or chronic hepatitis infection
   3. Any seizure disorder or evolving or unstable neurological condition
5. Anticipated cardiac surgery within 5-6 months after enrollment
6. Prior history of a suspected or actual acute life-threatening event
7. Receipt or intended use of palivizumab in the current enrollment season
8. Any known allergy or history of allergic reaction to any component of nirsevimab
9. Any known allergy or history of allergic reaction to immunoglobulin products, blood products, or other foreign proteins
10. Concurrent enrollment in another interventional study, or prior receipt of any investigational agent
11. Anticipated survival of less than 1 year at the time of informed consent
12. Any condition that, in the opinion of the investigator, would interfere with the evaluation of the investigational product or interpretation of study results
13. Children of employees of the Sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of all TEAEs, TESAEs, AESIs, and NOCDs | 360 days after the 2nd or last dose administered in the study
  The number and percentage of participants with TEAEs, TESAEs, AESIs, and NOCDs will be summarized by SOC and PT overall.
Study discontinuations prior to Day 151 post 2nd dose. | 360 days after the 2nd or last dose administered in the study
  The number and percentage of subject discontinuations will be summarized.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) - Nirsevimab serum concentrations | 360 days after the 2nd or last dose administered in the study
ADA - Occurrence of ADA to nirsevimab in serum | 360 days after the 2nd or last dose administered in the study
Anti-RSV neutralizing Ab - Anti-RSV neutralizing Ab levels (IU/mL) in serum | 360 days after the 2nd or last dose administered in the study

OTHER OUTCOMES:
MA-RSV LRTI - Occurrence of MA-LRTI (inpatient and outpatient) due to RT-PCR-confirmed RSV | through 150 and 360 days post 2nd dose
MA-RSV LRTI - Occurrence of hospitalizations due to RT-PCR-confirmed RSV | through 150 and 360 days post 2nd dose
Monitoring for RSV Resistance - Genotypic analysis of the F protein from collected RSV-positive respiratory secretion specimens | through 150 and 360 days post 2nd dose
Monitoring RSV Resistance to Nirsevimab - RSV novel variants will be phenotypically characterized for nirsevimab susceptibility | through 150 and 360 days post 2nd dose

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - Research Site, Bunkyō City
  - Research Site, Fuchu-shi
  - Research Site, Fukuoka
  - Research Site, Kitakyusyu-shi
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Nagasaki
  - Research Site, Saitama-shi
  - Research Site, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home